CLINICAL TRIAL: NCT03122509
Title: Phase II Study to Assess the Efficacy of Durvalumab (MEDI4736) and Tremelimumab Plus Radiotherapy or Ablation in Patients With Metastatic Colorectal Cancer
Brief Title: A Clinical Trial of Durvalumab and Tremelimumab, Administered With Radiation Therapy or Ablation in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: MedImmune LLC (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-139
Record Dates: First submitted 2017-04-18; First posted 2017-04-20 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Durvalumab; Tremelimumab; Radiation Therapy; Ablation; 17-139
MeSH Terms: conditions — Colorectal Neoplasms | interventions — durvalumab; tremelimumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This will be a Simon two-stage design, phase II study. It will be conducted to determine the efficacy and safety of (1) durvalumab and tremelimumab plus RT in subjects with metastatic CRC who are undergoing RT as standard therapy; and, (2) durvalumab and tremelimumab plus ablation in subjects with metastatic CRC who are undergoing ablation as standard therapy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- durvalumab and tremelimumab plus Radiotherapy (RT) (Experimental): Patients will receive 1500 mg durvalumab via IV infusion q4w for up to 4 doses/cycles and 75 mg tremelimumab via IV infusion q4w for up to 4 doses/cycles, and then continue 1500 mg durvalumab q4w starting on Week 16. Tremelimumab will be administered first. Durvalumab infusion will start approximately 1 hour after the end of tremelimumab infusion. The duration will be approximately 1 hour for each infusion. Radiotherapy (RT) will be performed using external beam ionizing radiation as standard therapy in accordance with institutional standard practice. RT will be initiated within 7 days after the first of durvalumab and tremelimumab.
  Interventions: Drug: durvalumab; Drug: tremelimumab; Radiation: Radiotherapy (RT)
- durvalumab and tremelimumab plus ablation (Experimental): Patients will receive 1500 mg durvalumab via IV infusion q4w for up to 4 doses/cycles and 75 mg tremelimumab via IV infusion q4w for up to 4 doses/cycles, and then continue 1500 mg durvalumab q4w starting on Week 16. Tremelimumab will be administered first. Durvalumab infusion will start approximately 1 hour after the end of tremelimumab infusion. The duration will be approximately 1 hour for each infusion. The ablation will be performed percutaneously under image guidance as standard therapy at the discretion of the interventional radiologist in accordance with institutional standard practice. Ablation will be performed within 7 days after the first of durvalumab and tremelimumab.
  Interventions: Drug: durvalumab; Drug: tremelimumab; Procedure: ablation

INTERVENTIONS:
Drug: durvalumab — 1500 mg durvalumab via IV infusion
  Other Names: (MEDI4736)
Drug: tremelimumab — 75 mg tremelimumab via IV infusion
Radiation: Radiotherapy (RT) — Radiotherapy (RT) will be performed using external beam ionizing radiation as standard therapy in accordance with institutional standard practice.
  Arms: durvalumab and tremelimumab plus Radiotherapy (RT)
Procedure: ablation — Ablation will be performed percutaneously under image guidance as standard therapy at the discretion of the interventional radiologist in accordance with institutional standard practice.
  Arms: durvalumab and tremelimumab plus ablation

SUMMARY:
The purpose of this study is to test the safety and effectiveness of two investigational drugs (drugs that are not currently approved by the FDA) given in combination with radiation therapy or ablation.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Histologically- or cytologically- confirmed CRC.
* Metastatic CRC.
* Subjects have received at least two standard chemotherapy regimens for which they would be considered eligible (at least one containing a 5-fluoropyrimidine), or systemic chemotherapy is not indicated in the setting of low volume metastatic disease.
* At least one tumor for which palliative RT is considered appropriate standard therapy (cohort 1); or, at least one tumor for which palliative ablation is considered appropriate standard therapy (cohort 2).
* At least one index lesion that will not undergo RT or ablation, and which is measurable based on RECIST 1.1.
* Be ≥ 18 years of age on day of signing informed consent.
* Consent for tumor biopsies (for patients enrolled in stage 1 only) and blood draws for research purposes (for all patients).
* Consent for use of available archived tissue and tumor obtained during a standard procedure, for research purposes.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: ≥60 years old and no menses for ≥ 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test within 2 weeks prior to starting treatment.
* Demonstrate adequate organ function as defined all screening labs should be performed within 4 weeks prior to treatment initiation.

  * Hemoglobin ≥ 8.0 g/dL
  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Serum creatinine ≤1.5 X upper limit of normal (ULN) OR
  * Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) OR
  * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases.

aCreatinine clearance should be calculated per institutional standard.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Chemotherapy, monoclonal antibody, targeted small molecule therapy, within 4 weeks prior to dose #1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent (excluding alopecia or toxicity not anticipated to interfere with planned treatment on study).
* Known or suspected MSI-H CRC.
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1, including anti-PD-1, anti-PD-L1, anti-CD137, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways, except for endocrinopathies and asymptomatic amylase/lipase.
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention per clinical discretion of the investigator prior to starting therapy.
* Concurrent active malignancy that requires systemic treatment.
* Known CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable without evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. The use of topical steroids is permitted.
* Active autoimmune disease requiring systemic immune suppressive treatment within the past 2 years. NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Has active, non-infectious pneumonitis.
* Active or prior documented inflammatory bowel disease.
* History of allogeneic organ transplant.
* Has an active infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active and untreated Hepatitis B (e.g., HBsAg reactive) or active Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab with the exceptions of premedication and intranasal, topical and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10mg/day of prednisone, or an equivalent corticosteroid.
* Hypersensitivity to durvalumab or tremelimumab, or any excipients on the formulation.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.
* QT interval corrected for heart rate (QTc) ≥ 470ms calculated from 1 electrocardiogram (ECG) using Fridericia's Correction.
* History of primary immunodeficiency.
* Known history of previous clinical diagnosis of tuberculosis.
* Subjects with uncontrolled seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Segal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab and Tremelimumab Plus Radiotherapy (RT): Patients will receive 1500 mg durvalumab via IV infusion q4w for up to 4 doses/cycles and 75 mg tremelimumab via IV infusion q4w for up to 4 doses/cycles, and then continue 1500 mg durvalumab q4w starting on Week 16. Tremelimumab will be administered first. Durvalumab infusion will start approximately 1 hour after the end of tremelimumab infusion. The duration will be approximately 1 hour for each infusion.
  RT will be initiated within 7 days after the first of durvalumab and tremelimumab.
- Durvalumab and Tremelimumab Plus Ablation: Patients will receive 1500 mg durvalumab via IV infusion q4w for up to 4 doses/cycles and 75 mg tremelimumab via IV infusion q4w for up to 4 doses/cycles, and then continue 1500 mg durvalumab q4w starting on Week 16. Tremelimumab will be administered first. Durvalumab infusion will start approximately 1 hour after the end of tremelimumab infusion. The duration will be approximately 1 hour for each infusion.
  Ablation will be performed within 7 days after the first of durvalumab and tremelimumab.
Period: Overall Study
Arm/Group | Durvalumab and Tremelimumab Plus Radiotherapy (RT) | Durvalumab and Tremelimumab Plus Ablation
Started | 25 | 0
Completed | 25 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were assigned to the Durvalumab and Tremelimumab + ablation arm.
Groups:
- Durvalumab and Tremelimumab Plus Radiotherapy (RT) or Ablation: Patients will receive 1500 mg durvalumab via IV infusion q4w for up to 4 doses/cycles and 75 mg tremelimumab via IV infusion q4w for up to 4 doses/cycles, and then continue 1500 mg durvalumab q4w starting on Week 16. Tremelimumab will be administered first. Durvalumab infusion will start approximately 1 hour after the end of tremelimumab infusion. The duration will be approximately 1 hour for each infusion.
  RT will be initiated within 7 days after the first of durvalumab and tremelimumab.
- Total: Total of all reporting groups
Arm/Group | Durvalumab and Tremelimumab Plus Radiotherapy (RT) or Ablation | Durvalumab and Tremelimumab Plus Ablation | Total
Number analyzed (Participants) | 25 | 0 | 25
Age, Continuous [Median (Full Range); unit: years] | 55 [26 to 78] |  | 55 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 |  | 12
  Male | 13 |  | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 24 |  | 24
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 4 |  | 4
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 19 |  | 19
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 |  | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: No participants were enrolled on the Durvalumab and Tremelimumab + ablation arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab and Tremelimumab Plus Radiotherapy (RT)
Number analyzed (Participants) | 25
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 3
  Progressive Disease | 19
  Unevaluable | 1

ADVERSE EVENTS:
Time Frame: 2 years
Description: No participants were assigned to the Durvalumab and Tremelimumab + ablation arm.
Arm/Group | Durvalumab and Tremelimumab Plus Radiotherapy (RT) or Ablation | Durvalumab and Tremelimumab Plus Ablation
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/0
Serious Adverse Events (participants affected / at risk) | 9/25 | 0/0
Other Adverse Events (participants affected / at risk) | 6/25 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab and Tremelimumab Plus Radiotherapy (RT) or Ablation (N=25) | Durvalumab and Tremelimumab Plus Ablation (N=0)
Biliary tract infection (Infections and infestations) | 1 | NA
Blood bilirubin increased (Investigations) | 1 | NA
Colitis (Gastrointestinal disorders) | 1 | NA
Enterocolitis infectious (Infections and infestations) | 1 | NA
Fever (General disorders) | 1 | NA
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | NA
Gen disorders & admin site conditions Other, spec (General disorders) | 1 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 1 | NA
Ileus (Gastrointestinal disorders) | 1 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Rectal hemorrhage (Gastrointestinal disorders) | 1 | NA
Sepsis (Infections and infestations) | 1 | NA
Upper respiratory infection (Infections and infestations) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab and Tremelimumab Plus Radiotherapy (RT) or Ablation (N=25) | Durvalumab and Tremelimumab Plus Ablation (N=0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 | NA
Alanine aminotransferase increased (Investigations) | 1 | NA
Aspartate aminotransferase increased (Investigations) | 1 | NA
Platelet count decreased (Investigations) | 1 | NA
Alkaline phosphatase increased (Investigations) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03122509/Prot_SAP_000.pdf